CLINICAL TRIAL: NCT06715475
Title: A Verification Study to Evaluate the Safety of Long-term Consumption of the Test Food: a Randomized, Placebo-controlled, Double-blind, Parallel-group Comparison Study
Brief Title: A Verification Study to Evaluate the Safety of Long-term Consumption of the Test Food
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Orthomedico Inc. (Other)
Collaborators: AOBA KASEI CO., LTD. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 04400-0006-06
Record Dates: First submitted 2024-11-22; First posted 2024-12-04 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Healthy Japanese
Keywords: Plasmalogen; Safety; Sleep condition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Plasmalogen (Active Comparator): Take 1 mg/day of plasmalogen
  Interventions: Dietary Supplement: Food containing plasmalogen
- Placebo (Placebo Comparator): Take 0 mg/day of plasmalogen
  Interventions: Dietary Supplement: Food not containing plasmalogen

INTERVENTIONS:
Dietary Supplement: Food containing plasmalogen — Take five capsules per day in the morning.
  Arms: Plasmalogen
Dietary Supplement: Food not containing plasmalogen — Take five capsules per day in the morning.
  Arms: Placebo

SUMMARY:
This clinical study aims to verify the safety of consumption of plasmalogen-containing food for 12 weeks in healthy Japanese. The study will also exploratory assess blood plasmalogen levels and the effects of plasmalogen-containing food on sleep.

DETAILED DESCRIPTION:
In this study, the investigators will confirm the safety of consumption of plasmalogen-containing food for 12 weeks in healthy Japanese. The investigators will also exploratory assess blood plasmalogen levels and the effect of plasmalogen-containing food on sleep conditions. The groups to be compared are plasmalogen-containing food and a placebo (plasmalogen-free food).

ELIGIBILITY:
Inclusion Criteria:

1. Japanese
2. Men or women
3. Adults
4. Healthy individuals

Exclusion Criteria:

1. Individuals who are undergoing medical treatment or have a medical history of malignant tumor, heart failure, or myocardial infarction
2. Individuals who have a pacemaker or an implantable cardioverter defibrillator (ICD)
3. Individuals who are currently undergoing treatment for any of the following chronic diseases: cardiac arrhythmia, liver disorder, chronic kidney disease, cerebrovascular disorder, rheumatic disease, diabetes mellitus, dyslipidemia, hypertension, or any other chronic diseases
4. Individuals who are undergoing medical treatment or have a medical history for any of the following diseases: mental disorder (such as depression), sleep apnea syndrome, hypersomnia, narcolepsy, insomnia, or valvular heart disease
5. Individuals who have habits of consuming foods or using devices to improve sleep
6. Individuals who have irregular sleeping habits due to lifestyle such as night shifts
7. Individuals who fall under the following sleeping conditions: sleeping in the same room with two or more people, living with preschool-aged children, living with individuals who require nursing care, or having their sleep potentially disturbed by the influence of others
8. Individuals who have nocturia two times or more
9. Individuals who usually drink to excess (average of more than about 20 g/day as absolute alcohol intake) {500 mL: a medium bottle of beer or about 1.5 cans of canned chu-hi, 180 mL: 1 go of sake or about 1.5 glasses of wine, 90 mL: half-go with shochu, 60 mL: a glass of whiskey brandy (double)}
10. Individuals who are taking "Foods for Specified Health Uses" or "Foods with Functional Claims"
11. Individuals who are taking medications (including herbal medicines) or supplements
12. Individuals who are allergic to medicines or foods related to the test product
13. Individuals who are pregnant, lactating, or planning to become pregnant during this study
14. Individuals who have been enrolled in other clinical studies within the last 28 days before the agreement to participate in this study or plan to participate in another study during this study
15. Individuals who are judged as ineligible to participate in this study by the physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-04-23 (Estimated); Study Completion 2025-04-23 (Estimated)

PRIMARY OUTCOMES:
Number of individuals who experienced adverse events | Intervention period (up to 12 weeks)
  An adverse event is defined as the "development of a new abnormality" or "worsening" in physical signs, symptoms, etc. that is clinically meaningful to the study participant during the study period, and the investigator will evaluate the relationship between the adverse event and the test product.

SECONDARY OUTCOMES:
Number of individuals whose values of blood test and urinalysis are outside the reference range after intervention despite within the reference range at Baseline (before intervention) | Week 6 and Week 12
  Count the number of individuals whose values of blood test items (white blood cell count, red blood cell count, hemoglobin level, hematocrit value, platelet count, aspartate transaminase, alanine transaminase, γ-glutamyltransferase, total bilirubin, total protein, urea nitrogen, creatinine, uric acid, sodium, potassium, chloride, serum amylase, total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, triglycerides, glucose, and hemoglobin A1c levels) and urinalysis items (urinary protein, glucose, pH, and occult blood) are outside the reference range after intervention (Week 6 and Week 12) despite within the reference range at Baseline.
The measured values of blood plasmalogen levels at Week 6 and Week 12 | Week 6 and Week 12
  This is one of the exploratory assessment items. Approximately 3 mL of venous blood will be collected from each study participant, and this sample will be analyzed.
The changes from baseline of blood plasmalogen levels at Week 6 and Week 12 | Baseline, Week 6, and Week 12
  This is one of the exploratory assessment items. Approximately 3 mL of venous blood will be collected from each study participant, and this sample will be analyzed.
Each questionnaire item in the St. Mary's Hospital Sleep Questionnaire (SMH) at Week 6 and Week 12 | Week 6 and Week 12
  These are one of the exploratory assessment items. The SMH is a self-administered tool to evaluate sleep over the past 24 hours. It includes questions with various response formats, such as yes/no answers, open-ended responses requiring specific time and time-of-day entries, and multiple-choice items with four or more options. Responses to the questions are reviewed individually.

CONTACTS AND LOCATIONS:
Overall Officials: Tsuyoshi Takara, MD, Study Chair — Medical Corporation Seishinkai, Takara Clinic
Locations (2):
- Japan (2):
  - Nerima Medical Association Minami-machi Clinic, Nerima-ku, Tokyo
  - Medical Corporation Seishinkai, Takara Clinic, Shinagawa-ku, Tokyo

IPD SHARING:
Plan to Share IPD: No
Data sharing will be discussed among the research affiliates after the study is completed.